CLINICAL TRIAL: NCT03738761
Title: Fixed-Dose Combination of Perindopril/Amlodipine (Amlessa®) and Fixed-Dose Combination of Perindopril/Indapamide /Amlodipine (Co-Amlessa®) - Contribution to Management in Newly Diagnosed and Uncontrolled Hypertensive Patients
Brief Title: Management of Newly Diagnosed and Uncontrolled Hypertension With Fixed-Dose Combination of Perindopril/Amlodipine and Perindopril/Indapamide/Amlodipine
Acronym: PRECIOUS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: KRKA (Industry)
Collaborators: Clinres Farmacija d.o.o. (Industry); University Medical Centre Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: KCT 06/2017; 2017-001596-23 (EudraCT Number)
Record Dates: First submitted 2018-10-30; First posted 2018-11-13 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2019-09

CONDITIONS: Hypertension
Keywords: Hypertension; Blood pressure control; Fixed-dose combination antihypertensives; Ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Treatment is started at Visit 1 with Amlessa® 4mg/5mg (Amlessa® Arm) or Co-Amlessa® 4mg/1,25mg/5mg (Co-Amlessa® Arm) for 4 weeks.
  At each of the three follow-up visits (at week 4, week 8 and week 12) patient BP is assessed and if normal office blood pressure was achieved, the treatment with the study medication prescribed for the previous treatment period is continued. If normal office blood pressure was not achieved at any of the follow-up visits (week 4, week 8 and week 12), Amlessa® or Co-Amlessa® strength is increased in accordance with the below sequence.
  Amlessa® Arm Amlessa® 4mg/5mg (initial therapy) - Amlessa® 8mg/5mg - Amlessa® 8mg/10mg - Co-Amlessa® 8mg/2,5mg/10mg
  Co-Amlessa® Arm Co-Amlessa® 4mg/1,25mg/5mg - Co-Amlessa® 8mg/2,5mg/5mg - Co-Amlessa® 8mg/2,5mg/10mg - end of study no further escalation of study medication dosage
  Normal office BP is defined as SBP < 140 mmHg and DBP < 90 mmHg; patients with type 2 diabetes mellitus: SBP < 140 mmHg and DBP < 85 mmHg.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amlessa® Arm (Experimental): Patients allocated to treatment with Amlessa® (starting FDC of perindopril 4mg/amlodipine 5mg) according to their previous antihypertensive therapy and as described in the protocol inclusion criteria.
  Interventions: Drug: Amlessa®; Drug: Co-Amlessa®
- Co-Amlessa® Arm (Experimental): Patients allocated to treatment with Co-Amlessa® (starting FDC perindopril 4mg/indapamide 2,5mg/amlodipine 5mg) according to their previous antihypertensive therapy and as described in the protocol inclusion criteria. Patients on previous perindopril and amlodipine therapy will be automatically assigned to Co-Amlessa® arm.
  Interventions: Drug: Co-Amlessa®

INTERVENTIONS:
Drug: Amlessa® — Fixed-dose combination (FDC) of perindopril/amlodipine, tablets. Strengths: 4mg/5 mg, 8mg/5 mg, 8mg/10 mg.
  Arms: Amlessa® Arm
Drug: Co-Amlessa® — Fixed-dose combination (FDC) of perindopril/indapamide/amlodipine, tablets. Strengths: 4mg/1.25 mg/5 mg, 8mg/2.5 mg/5 mg, 8mg/2.5 mg/10 mg.

SUMMARY:
PRECIOUS Study aims to evaluate the efficacy and safety of therapy with fixed-dose combination (FDC) of perindopril/amlodipine (Amlessa®) and FDC of perindopril/indapamide/amlodipine (Co-Amlessa®) on blood pressure reduction in both previously untreated patients and patients with previous antihypertensive therapy.

Adult patients with AH who are treatment-naïve with systolic blood pressure (SBP) from 150 mmHg or higher AND/OR diastolic blood pressure (DBP) from 95 mmHg or higher (SBP ≥ 150 mm AND/OR DBP ≥ 90 mmHg for patients with type 2 diabetes mellitus ) and uncontrolled patients on mono, dual or triple antihypertensive therapy with systolic blood pressure (SBP) from 140 mmHg or higher AND/OR diastolic blood pressure (DBP) from 90 mmHg or higher (SBP ≥ 140 AND/OR DBP ≥ 85 mmHg for patients with type 2 diabetes mellitus) will be invited to participate in this study.

During 16-week trial, seven study visits are planned. At first study visit physical examination, medical history, BP measurement, electrocardiogram (ECG), laboratory analysis and of Ambulatory Blood Pressure Measurement (ABPM) will be performed. Based on their previous antihypertensive therapy, patients will receive to treatment with either Amlessa® or Co-Amlessa® for the duration of 16 weeks and blood pressure measurements, laboratory investigations and patient interviews will be performed at study follow-up visits to assess the treatment efficacy (proportion of patients reaching normal office blood pressure after 16 weeks of treatment) and safety.

DETAILED DESCRIPTION:
PRECIOUS study is an interventional, open-label, prospective, international, multi-centre, Phase IV clinical trial (Phase III for countries without marketing authorisation for Co-Amlessa®).

The purpose of the study is to establish the efficacy and safety of fixed-dose combination (FDC) of perindopril/amlodipine (Amlessa®) and FDC of perindopril/indapamide/amlodipine (Co-Amlessa®) in wide populations of newly diagnosed and uncontrolled patients with arterial hypertension (AH) with special focus on effective continuous 24-hour blood pressure (BP) control. The purpose is also to establish the correlation between 24-hour central and peripheral BP.

Perindopril, indapamide and amlodipine are well known and extensively studied antihypertensive monotherapies. Clinical data and safety analyses provided are substantial body of evidence that perindopril, indapamide and amlodipine, which have been used for more than 15 years, are safe and well tolerated drugs. Perindopril, indapamide and amlodipine have complementary actions in reducing BP. Combining perindopril and amlodipine or perindopril, indapamide and amlodipine could improve adherence in uncontrolled hypertensive patients. Namely the combinations would reduce the number of tablets to be taken by patient and thus simplify the treatment regimen and are therefore expected to facilitate long-term adherence to antihypertensive therapy, which justifies their use. Both combinations could also improve safety profile which would be beneficial from the tolerability point of view. Namely, when calcium channel blockers (CCB) and angiotensin converting enzyme inhibitors (ACEI) are used in combination, there is a potential for lower incidence of peripheral oedema caused by CCB. Similarly, the incidence of ACEI-associated cough is attenuated by CCBs, including amlodipine.

This study aims evaluate the effect of therapy with Amlessa® and Co-Amlessa® on the blood pressure reduction in patients with essential arterial hypertension (AH) who are naïve with systolic blood pressure (SBP) from 150 mmHg or higher AND/OR diastolic blood pressure (DBP) from 95 mmHg or higher, (SBP ≥ 150 AND/OR DBP ≥ 90 mmHg for patients with type 2 diabetes mellitus) and in uncontrolled patients on mono, dual or triple antihypertensive with SBP from 140 mmHg or higher AND/OR DBP from 90 mmHg or higher (SBP ≥ 140 AND/OR DBP ≥ 85 mmHg for patients with type 2 diabetes mellitus). An objective of this trial is also to evaluate the safety of therapy with Amlessa® and Co-Amlessa® according to the frequency and severity of AR in patients with essential AH. Overall 510 patients are planned to conclude the assessment and to be analysed. In per-protocol analysis 450 patients are expected. In order to allow for the estimated drop-out rate, up to 570 patients are expected to be screened.

All patients start with an initial screening which is performed one day before visit 1 to verify eligibility. After inform consent signature and before therapy is allocated complete medical history, physical examination with measurements of heart rate (HR), body weight and height, lipid measurements and laboratory analysis including pregnancy test, BP, ambulatory blood pressure measurement (ABPM) and electrocardiogram (ECG) are performed. Patients take the last doses of previous AH therapy on the day of the screening visit. At Visit 1 (day 0) the data from ABPM device is collected (average BP, central BP, HR, pulse wave velocity [PWV] and Aortic augmentation index). BP and HR measurements are repeated. Based on data gathered from all previous examinations on visit -1 and visit 1 investigator verifies patient's eligibility. Patients will not be randomized to treatment. All eligible patients are assigned to start receiving any of the two study medication (Amlessa® and Co-Amlessa®) according to their previous antihypertensive therapy and as described in the protocol inclusion criteria. Patients on previous perindopril and amlodipine therapy will be automatically assigned to Co-Amlessa® group. Patient starts taking the study medication on day of the visit 1 (day 0).

The total active treatment duration is 16 weeks, with maximal allowed prolongation of 3 additional days per each of the four treatment periods due to possible unpredicted causes for delay in the follow-up visits. The whole trial treatment schedule was determined on the basis of published pharmacological data for all active substances in study medications. During the active treatment period each patient orally consumes one unit of assigned study medication once daily, at about the same time each day (± 3 hours), preferably in the morning and before a meal.

At visit 2, on day 28 of the treatment period, BP, HR measurements, safety assessing laboratory investigations (serum creatinine, serum potassium, ALT, AST, GammaGT) are repeated. Patient's compliance is assessed and safety assessment is carried out by the interview. After the control of patient status the decision is made to maintain the treatment if sufficient (normal office BP was reached) or to change the treatment in accordance with protocol treatment model. Normal office BP is defined as SBP < 140 mmHg and DBP < 90 mmHg; patients with type 2 diabetes mellitus: SBP < 140 mmHg and DBP < 85 mmHg.

At Visit 3 on day 56 of the active treatment period, BP, HR measurements measurements, lipid measurements and safety assessing laboratory investigations (serum creatinine, serum potassium, ALT, AST, GammaGT) are repeated. Patient's compliance is assessed and safety assessment is carried out by the interview. After the control of patient status the decision is made to maintain the treatment if sufficient (normal office BP was reached) or to change the treatment in accordance with protocol treatment model. Normal office BP is defined as SBP < 140 mmHg and DBP < 90 mmHg; patients with type 2 diabetes mellitus: SBP < 140 mmHg and DBP < 85 mmHg.

At Visit 4 on day 84 of the active treatment period, BP, HR measurements measurements are repeated. Patient's compliance is assessed and safety assessment is carried out by the interview. After the control of patient status the decision is made to maintain the treatment if sufficient (normal office BP was reached) or to change the treatment in accordance with protocol treatment model. Normal office BP is defined as SBP < 140 mmHg and DBP < 90 mmHg; patients with type 2 diabetes mellitus: SBP < 140 mmHg and DBP < 85 mmHg.

At Visit -5 on day 111, ABPM device is installed. Blood samples are taken, to provide the results of laboratory analysis the next day on visit 5 (final visit). At Visit 5 on day 112, the final efficacy and safety evaluation are carried out including patient's adherence. Physical examination with BP, PWV and HR measurements, lipid measurements, laboratory analysis and ABPM are performed. ABPM device is removed on the same day and the data from device is collected (average BP, central BP, HR, PWV and Aortic augmentation index). Completion of all the procedures at Visit 5 determines the end of the patient's involvement in this clinical trial. After this, patient's further antihypertensive regimen is left to the discretion of the investigator.

Once enrolled, patients can be excluded before the protocol defined end of therapy due to patients decision or loss-to-follow-up, patient non-compliance or safety issues as defined in the study protocol. Concomitant therapy with other drugs is avoided in this study, if possible.

The primary efficacy endpoint is the responder rate at final visit. Precisely, this is defined to be the proportion of patients reaching normal blood pressure at Visit 5 (after 16 weeks). Normal office BP is defined as SBP < 140 mmHg and DBP < 90 mmHg; patients with type 2 diabetes mellitus: SBP < 140 mmHg and DBP < 85 mmHg. It will be assessed with the two-sided ("equal-tails") Clopper-Pearson exact 95%-confidence interval for a population proportion.

This trial is going to be conducted in compliance with the approved protocol and in accordance with the principles of Good Clinical Practice (GCP) with its corresponding Directives and Declaration of Helsinki. Data management is carried out by the sponsor according to the data management plan, sponsor's standard operating procedures (SOPs) and GCP. Data to be collected according to the study protocol (and amendments, if any) will be recorded in electronic case report forms (eCRF).

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with essential arterial hypertension.*
* Men and women aged ≥ 18 years
* Written informed consent
* Ability to adhere to study protocol

Additional inclusion criteria for Amlessa®*

Patients with essential arterial hypertension:

* Naïve patients with systolic blood pressure (SBP) from 150 mmHg or higher AND/OR diastolic blood pressure (DBP) from 95 mmHg or higher (SBP ≥ 150 AND/OR DBP ≥ 90 mmHg for patients with type 2 diabetes mellitus)
* Uncontrolled patients on antihypertensive monotherapy with SBP from 140 mmHg or higher AND/OR DBP from 90 mmHg or higher (SBP ≥ 140 AND/OR DBP ≥ 85 mmHg for patients with type 2 diabetes mellitus).
* Uncontrolled patients on dual antihypertensive therapy (either in monoforms or FDC) with SBP from 140 mmHg or higher AND/OR DBP from 90 mmHg or higher (SBP ≥ 140 AND/OR DBP ≥ 85 mmHg for patients with type 2 diabetes mellitus).

Additional inclusion criteria for Co-Amlessa®*

Patients with essential arterial hypertension (AH):

* Uncontrolled patients on dual antihypertensive therapy (either in monoforms or FDC, including perindopril+amlodipine combination) with SBP from 140 mmHg or higher AND/OR DBP from 90 mmHg or higher (SBP ≥ 140 AND/OR DBP ≥ 85 mmHg for patients with type 2 diabetes mellitus).
* Uncontrolled patients on triple antihypertensive therapy (either in monoforms or FDC) with SBP from 140 mmHg or higher AND/OR DBP from 90 mmHg or higher (SBP ≥ 140 AND/OR DBP ≥ 85 mmHg for patients with type 2 diabetes mellitus).

EXCLUSION CRITERIA:

* History of adverse reactions or hypersensitivity associated with the use of the active substances, or any other components of the Investigational medicinal products (IMPs) used in the trial.
* Hereditary/idiopathic angioedema.
* Known secondary AH (e.g. pheochromocytoma, primary aldosteronism, renal artery stenosis).
* Office measured Systolic blood pressure ≥200 mmHg.
* Unstable angina pectoris.
* Acute heart failure and heart failure New York Heart Association (NYHA) Class IV.
* Antihypertensive drugs used for other indication than AH (e.g. tachyarrhythmia, glaucoma) less than 3 months before the study or in changed dosages less than 3 months before the study.
* Severe liver impairment OR biliary cirrhosis OR cholestasis OR hepatic encephalopathy.
* Renal dysfunction - glomerular filtration rate (GFR) <60 ml/min, bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, patients with only 1 kidney, or post-renal transplant patients, dialysis patients.
* Any of the following clinically relevant laboratory or ECG findings:

  * significant anaemia with haemoglobin less than 100 g/l
  * serum aspartate transaminase (AST) and/or alanine aminotransferase (ALT) and/or alkaline phosphatase (ALP) and/or gamma-glutamyltransferase (GGT) of more than 3 x upper limit of normal (ULN)
  * hyperkalaemia (serum potassium of more than 5 mmol/l)
  * A-V block grade 2 or 3
  * ECG signs of acute ischemia
* Concurrent therapy with:

  * aliskiren-containing products (in patients with diabetes mellitus or renal impairment)
  * Other antihypertensive drugs or other medications that may cause hypotension: exception are antihypertensive drugs used for other indication than AH (e.g. tachyarrhythmia, glaucoma) introduced more than 3 months before the study or in changed dosages more than 3 months before the study
  * Drugs that may produce an increase in blood pressure: systemic corticosteroids, hormonal medications (chronically used oral contraceptives are allowed), adrenergic receptor agonists, cyclosporine, erythropoietin, migraine medications such as triptans and ergotamines
  * Agents with important interactions with perindopril or to any other ACE inhibitor, to indapamide or to any other sulphonamides, to amlodipine or to dihydropyridine derivatives: lithium, estramustine
  * Agents that may interfere with amlodipine hepatic metabolism (CYP3A4): protease inhibitors, rifampicin, macrolides like erythromycin or clarithromycin, azole antifungals like ketoconazole and itraconazole, Hypericum perforatum.
  * Medications contraindicated in uncontrolled arterial hypertension: anticoagulants, thrombolytics.
* Bradycardia with heart rate less than 50/min.
* Female patients who are pregnant, planning to become pregnant.
* Breastfeeding female patients.
* Any significant acute condition (severe infection, exacerbation or uncontrolled phase of a chronic disease, major trauma, major surgery) within 30 days prior to screening visit.
* Pathological clinical states (e.g. malignant diseases, excessive alcohol consumption, drug abuse or drug addiction, psychiatric conditions) or any life-threatening illness.
* Patients currently participating in another clinical trial.
* Patient's refusal to participate with the investigator.
* Normal average 24-hour SBP and DBP obtained by Ambulatory Blood Pressure Measurement (ABPM) device (<130/80 mmHg) at baseline.
* Severe orthostatic hypotension.
* Patients to whom β-blocker therapy cannot be discontinued in one day.
* Previous or current therapy with perindopril and amlodipine and indapamide taken taken concomitantly all together as 3 separate tablets or as a fixed-dose combination.
* In Amlessa arm patients on previous or current therapy with perindopril and amlodipine taken concomitantly all together as 2 separate tablets or as a fixed-dose combination. (this exclusion criterion does not apply to Co-Amlessa arm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2019-09-27 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic blood pressure at Week 16 | 16 weeks
  Responder rate at end of study (week 16): proportion of patients reaching office normal blood pressure defined as SBP < 140 mmHg and DBP < 90 mmHg (patients with type 2 diabetes mellitus: SBP < 140 mmHg and DBP < 85 mmHg). BP is measured using a validated automated BP-measuring device.

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure at Week 4, Week 8 and Week 12 | 12 Weeks
  Responder rate at first, second and third study follow-up visits (week 4, week 8 and week 12): proportion of patients reaching office normal blood pressure defined as SBP < 140 mmHg and DBP < 90 mmHg (patients with type 2 diabetes mellitus: SBP < 140 mmHg and DBP < 85 mmHg). BP is measured using a validated automated BP-measuring device.
Mean absolute and relative change in Systolic and diastolic blood pressure from baseline to Week 4, Week 8, Week 12 and Week 16 | 16 weeks
  Mean absolute and relative change from baseline in office SBP and DBP after 4, 8, 12 and 16 weeks (Visit 2, 3, 4, 5). BP is measured using a validated automated BP-measuring device.
Average 24-hour blood pressure at Week 16 | 16 weeks
  Proportion of patients reaching normal average 24h SBP and DBP (<130/80 mmHg) at study end (Week 16). Measurements are obtained with Ambulatory Blood Pressure Measuring (ABPM) device.
Average awake time blood pressure at Week 16 | 16 weeks
  Proportion of patients reaching normal average awake time SBP and DBP (<135/85 mmHg) at study end (Week 16). Measurements are obtained with Ambulatory Blood Pressure Measuring (ABPM) device.
Average sleep time blood pressure at Week 16 | 16 weeks
  Proportion of patients reaching normal average sleep time SBP and DBP (<120/70 mmHg) at study end (Week 16). Measurements are obtained with Ambulatory Blood Pressure Measuring (ABPM) device.
Mean absolute and relative change in average 24-hour blood pressure from baseline to Week 16 | 16 weeks
  Mean absolute and relative change from baseline to 16 weeks in average 24-hour SBP and DBP obtained with Ambulatory Blood Pressure Measuring (ABPM) device.
Mean absolute and relative change in average awake time blood pressure from baseline to Week 16 | 16 weeks
  Mean absolute and relative change from baseline to 16 weeks in average awake time SBP and DBP obtained with Ambulatory Blood Pressure Measuring (ABPM) device.
Mean absolute and relative change in average sleep time blood pressure from baseline to Week 16 | 16 weeks
  Mean absolute and relative change from baseline to 16 weeks in average sleep time SBP and DBP obtained with Ambulatory Blood Pressure Measuring (ABPM) device.
Reduction of office SBP of at least 20 mmHg or DBP of at least 10 mmHg from baseline to 16 weeks | 16 weeks
  Proportion of patients reaching a reduction of office SBP by at least 20 mmHg or DBP by at least 10 mmHg from baseline after 16 weeks. BP is measured using a validated automated BP-measuring device.
Central (systolic) blood pressure at Week 16 | 16 weeks
  Proportion of patients with a reduction of central (systolic) blood pressure (obtained by 24-hour ABPM device measurement) below 120 mmHg at end of study (week 16).
Change in Pulse wave velocity (PWV) from baseline to Week 16 | 16 weeks
  Proportion of patients reaching a reduction of PWV (obtained by 24-hour ABPM device measurement) of at least 0,5 m/s from baseline to study end (week 16).
Change in SBP and DBP variability from baseline to Week 16 | 16 weeks
  Proportion of patients reaching a reduction of SBP and DBP variability expressed as reduction of day-night standard deviation (SDdn) of at least 0.5 and that of average real variability (ARV) of at least 0.5 at study end (week 16). Measurements are obtained with ABPM device.

OTHER OUTCOMES:
Change in serum total cholesterol from baseline to end of study (Week 16) | 16 weeks
  Mean absolute and relative change from baseline to week 16 in total serum cholesterol concentration (obtained by laboratory blood test) in patients with concomitant rosuvastatin therapy.
Change in HDL-C from baseline to end of study (week 16) | 16 weeks
  Mean absolute and relative change from baseline to week 16 in high-density lipoprotein-cholesterol (HDL-C) serum concentration (obtained by laboratory blood test) in patients with concomitant rosuvastatin therapy.
Change in LDL-C from baseline to end of study (week 16) | 16 weeks
  Mean absolute and relative change from baseline to week 16 in low-density lipoprotein-cholesterol (LDL-C) serum concentration (obtained by laboratory blood test) in patients with concomitant rosuvastatin therapy.
Change in triglycerides from baseline to end of study (week 16) | 16 weeks
  Mean absolute and relative change from baseline to week 16 in triglycerides serum concentration (obtained by laboratory blood test) in patients with concomitant rosuvastatin therapy.
Change in AST from baseline to end of study (week 16) | 16 weeks
  Mean absolute and relative changes above normal limit values from baseline to end of study value (week 16) in serum Aspartate transaminase (AST) concentration obtained by laboratory blood test.
Change in ALT from baseline to end of study (week 16) | 16 weeks
  Mean absolute and relative changes above normal limit values from baseline to end of study value (week 16) in serum Alanine transaminase (ALT) concentration obtained by laboratory blood test.
Change in GGT from baseline to end of study (week 16) | 16 weeks
  Mean absolute and relative changes above normal limit values from baseline to end of study value (week 16) in serum gamma-glutamyl transferase (GGT) concentration obtained by laboratory blood test.
Change in Serum Creatinine from baseline to end of study (week 16) | 16 weeks
  Mean absolute and relative changes above normal limit values from baseline to end of study value (week 16) in Serum Creatinine concentration obtained by laboratory blood test.
Change in Serum Potassium from baseline to end of study (week 16) | 16 weeks
  Mean absolute and relative changes above normal limit values from baseline to end of study value (week 16) in Serum Potassium concentration obtained by laboratory blood test.
Incidence of adverse drug reactions from date of screening until study end (16 weeks) | 16 weeks
  Incidence of adverse drug reactions from date of screening until study end (16 weeks). A number/percentage of patients unable to finish active treatment periods due to clinically significant adverse reaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jana Brguljan Hitij, Principal Investigator — University Medical Centre Ljubljana Hospital dr. Peter Držaj
Locations (34):
- Armenia (2):
  - Unimed medical center, Abovyan
  - Center of Preventive Cardiology, Yerevan
- Croatia (7):
  - Thalassotherapia Opatija, Specijalna bolnica za medicinsku rehabilitaciju, bolesti srca, pluća i reumatizma, Klinika za liječenje, rehabilitaciju i prevenciju bolesti srca i krvnih žila, Opatija
  - KBC Rijeka - Sušak, Klinika za internu medicinu, Zavod za nefrologiju, dijalizu i transplantaciju bubrega, Rijeka
  - KB Merkur, Klinika za unutarnje bolesti, Zavod za kardiologiju, Zagreb
  - KBC Sestre milosrdnice, Klinika za bolesti srca i krvnih žila, Zavod za bolesti krvnih žila, Zagreb
  - KBC Zagreb, Klinika za bolesti srca i krvnih žila, Zagreb
  - KBC Zagreb, Klinika za unutarnje bolesti, Zavod za nefrologiju, arterijsku hipertenziju, dijalizu i transplantaciju, Zagreb
  - Poliklinika za prevenciju kardiovaskularnih bolesti i rehabilitaciju SRČANA, Zagreb
- Hungary (3):
  - Biatros Kft., Biatorbágy
  - General practitioner office, Budapest
  - AD SANITATEM Bt., Pilisvörösvár
- Poland (8):
  - Przychodnia Kardiologiczna w Zespole Przychodni Specjalistycznych DIAB-END-COR, Krakow
  - Niepubliczny Zakład Opieki Zdrowotnej Neuromed M.i M. Nastaj Spółka Partnerska, Lublin
  - Poradnia Kardiologiczna, Nowodworskie Centrum Medyczne, Nowy Dwór Mazowiecki
  - Poradnia Kardiologiczna Samodzielnego Publicznego Zespołu Zakładów Opieki Zdrowotnej im. Marszałka Józefa Piłsudskiego w Płońsku, Płońsk
  - Poradnia Kardiologiczna w Niepublicznym Zakładzie Opieki Zdrowotnej Euro-Klinika Sp. z o.o. w Siemianowicach Śląskich, Siemianowice Śląskie
  - Poradnia internistyczno-kardiologiczna w Niepublicznym Zakładzie Opieki Zdrowotnej AURUM, Warsaw
  - Poradnia Kardiologiczna w Przychodni Rejonowej - Specjalistycznej (III) Samodzielnego Zespołu Publicznych Zakładów Lecznictwa Otwartego Warszawa - Ochota, Warsaw
  - Przychodnia ACTIV-MED., Warsaw
- Russia (5):
  - Federal State Budgetary Scientific Institution "Scientific Research Institute of Complex Problems of Cardiovascular Diseases", Kemerovo
  - Federal State budget organization National medical research center of cardiology of the Ministry of healthcare of the Russian Federation, Moscow
  - State Budgetary Institution of Healthcare of Moscow "City Clinical Hospital № 29 named after N.E. Bauman of Department of Healthcare of Moscow city" (SBIH "CCH № 29 Bauman"), Moscow
  - Federal State Budgetary Institution "V.A. Almazov National Medical Research Center" of the Ministry of Health of the Russian Federation (V.A. Almazov NMRC), Saint Petersburg
  - Federal State Budgetary Educational Institution Higher Education "Volgograd State Medical University" of the Ministry of Healthcare of the Russian Federation (FSBEI HE VolgSMU MOH Russia), Volgograd
- Serbia (4):
  - KBC Dragiša Mišović, Belgrade
  - Klinički centar Srbije, Belgrade
  - Inštitut za kardiovaskularne bolesti Vojvodine, Kamenitz
  - Klinički centar Niš, Niš
- Slovenia (5):
  - Univerzitetna klinika za pljučne bolezni in alergijo Golnik, Golnik
  - Splošna bolnišnica Jesenice, Jesenice
  - Ordinacija interne medicine Verboten Kopriva Renata, Litija
  - MC Medicor, d. d., Ljubljana
  - Intermed, d. o. o., Maribor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waeber B, Feihl F, Ruilope LM. Fixed-dose combinations as initial therapy for hypertension: a review of approved agents and a guide to patient selection. Drugs. 2009;69(13):1761-76. doi: 10.2165/11316710-000000000-00000. PMID 19719332
- [Background] Whitworth JA; World Health Organization, International Society of Hypertension Writing Group. 2003 World Health Organization (WHO)/International Society of Hypertension (ISH) statement on management of hypertension. J Hypertens. 2003 Nov;21(11):1983-92. doi: 10.1097/00004872-200311000-00002. PMID 14597836
- [Background] Schmieder RE. The role of fixed-dose combination therapy with drugs that target the renin-angiotensin system in the hypertension paradigm. Clin Exp Hypertens. 2010 Jan;32(1):35-42. doi: 10.3109/10641960902960532. PMID 20144071
- [Background] Degaute JP, Leeman M, Desche P. Long-term acceptability of perindopril: European multicenter trial on 856 patients. Am J Med. 1992 Apr 27;92(4B):84S-90S. doi: 10.1016/0002-9343(92)90154-4. PMID 1580287
- [Background] Speirs C, Wagniart F, Poggi L. Perindopril postmarketing surveillance: a 12 month study in 47,351 hypertensive patients. Br J Clin Pharmacol. 1998 Jul;46(1):63-70. doi: 10.1046/j.1365-2125.1998.00031.x. PMID 9690951
- [Background] Cohn JN, Julius S, Neutel J, Weber M, Turlapaty P, Shen Y, Dong V, Batchelor A, Guo W, Lagast H. Clinical experience with perindopril in African-American hypertensive patients: a large United States community trial. Am J Hypertens. 2004 Feb;17(2):134-8. doi: 10.1016/j.amjhyper.2003.09.017. PMID 14751655
- [Background] Guo W, Turlapaty P, Shen Y, Dong V, Batchelor A, Barlow D, Lagast H. Clinical experience with perindopril in patients nonresponsive to previous antihypertensive therapy: a large US community trial. Am J Ther. 2004 May-Jun;11(3):199-205. doi: 10.1097/00045391-200405000-00008. PMID 15133535
- [Background] Kuwajima I, Fujisawa A, Mitani K, Suzuki Y, Kuramoto K. Effect of perindopril on 24-hour blood pressure levels and hemodynamic responses to physical and mental stress in elderly hypertensive patients. Clin Ther. 1994 Nov-Dec;16(6):962-71. PMID 7697693
- [Background] Suraniti S, Berrut G, Marre M, Fressinaud P. Antihypertensive efficacy and acceptability of perindopril in elderly hypertensive patients. Am J Cardiol. 1993 Jun 24;71(17):28E-31E. doi: 10.1016/0002-9149(93)90949-d. PMID 8328364
- [Background] Leenen FH, Tanner J, McNally CF. Antihypertensive efficacy of the ACE-inhibitor perindopril in the elderly. J Hum Hypertens. 2000 May;14(5):321-5. doi: 10.1038/sj.jhh.1001004. PMID 10822319
- [Background] Davis BR, Cutler JA, Gordon DJ, Furberg CD, Wright JT Jr, Cushman WC, Grimm RH, LaRosa J, Whelton PK, Perry HM, Alderman MH, Ford CE, Oparil S, Francis C, Proschan M, Pressel S, Black HR, Hawkins CM. Rationale and design for the Antihypertensive and Lipid Lowering Treatment to Prevent Heart Attack Trial (ALLHAT). ALLHAT Research Group. Am J Hypertens. 1996 Apr;9(4 Pt 1):342-60. doi: 10.1016/0895-7061(96)00037-4. PMID 8722437
- [Background] Zannad F, Bernaud CM, Fay R. Double-blind, randomized, multicentre comparison of the effects of amlodipine and perindopril on 24 h therapeutic coverage and beyond in patients with mild to moderate hypertension. General Physicians Investigators' Group. J Hypertens. 1999 Jan;17(1):137-46. doi: 10.1097/00004872-199917010-00020. PMID 10100105
- [Background] Oparil S, Barr E, Elkins M, Liss C, Vrecenak A, Edelman J. Efficacy, tolerability, and effects on quality of life of losartan, alone or with hydrochlorothiazide, versus amlodipine, alone or with hydrochlorothiazide, in patients with essential hypertension. Clin Ther. 1996 Jul-Aug;18(4):608-25. doi: 10.1016/s0149-2918(96)80212-8. PMID 8879890
- [Background] Neaton JD, Grimm RH Jr, Prineas RJ, Stamler J, Grandits GA, Elmer PJ, Cutler JA, Flack JM, Schoenberger JA, McDonald R, et al. Treatment of Mild Hypertension Study. Final results. Treatment of Mild Hypertension Study Research Group. JAMA. 1993 Aug 11;270(6):713-24. PMID 8336373
- [Background] Lefebvre J, Poirier L, Archambault F, Jewell D, Reed CV, Lacourciere Y. Comparative effects of felodipine ER, amlodipine and nifedipine GITS on 24 h blood pressure control and trough to peak ratios in mild to moderate ambulatory hypertension: a forced titration study. Can J Cardiol. 1998 May;14(5):682-8. PMID 9627524
- [Background] Emeriau JP, Knauf H, Pujadas JO, Calvo-Gomez C, Abate G, Leonetti G, Chastang C; European Study Investigators. A comparison of indapamide SR 1.5 mg with both amlodipine 5 mg and hydrochlorothiazide 25 mg in elderly hypertensive patients: a randomized double-blind controlled study. J Hypertens. 2001 Feb;19(2):343-50. doi: 10.1097/00004872-200102000-00023. PMID 11212979
- [Background] Frishman WH, Brobyn R, Brown RD, Johnson BF, Reeves RL, Wombolt DG. Amlodipine versus atenolol in essential hypertension. Am J Cardiol. 1994 Jan 27;73(3):50A-54A. doi: 10.1016/0002-9149(94)90275-5. PMID 8310977
- [Background] Osterloh I. The safety of amlodipine. Am Heart J. 1989 Nov;118(5 Pt 2):1114-9; discussion 1119-20. doi: 10.1016/0002-8703(89)90838-7. PMID 2573265
- [Background] Lau CP, Cheung BM. Relative efficacy and tolerability of lacidipine and amlodipine in patients with mild-to-moderate hypertension: a randomized double-blind study. J Cardiovasc Pharmacol. 1996 Aug;28(2):328-31. doi: 10.1097/00005344-199608000-00021. PMID 8856491
- [Background] Haria M, Wagstaff AJ. Amlodipine. A reappraisal of its pharmacological properties and therapeutic use in cardiovascular disease. Drugs. 1995 Sep;50(3):560-86. doi: 10.2165/00003495-199550030-00009. PMID 8521773
- [Background] Lorimer AR, Lyons D, Fowler G, Petrie JC, Rothman MT. Differences between amlodipine and lisinopril in control of clinic and twenty-four hour ambulatory blood pressures. J Hum Hypertens. 1998 Jun;12(6):411-6. doi: 10.1038/sj.jhh.1000620. PMID 9705044
- [Background] Corea L, Cardoni O, Fogari R, Innocenti P, Porcellati C, Provvidenza M, Meilenbrock S, Sullivan J, Bodin F. Valsartan, a new angiotensin II antagonist for the treatment of essential hypertension: a comparative study of the efficacy and safety against amlodipine. Clin Pharmacol Ther. 1996 Sep;60(3):341-6. doi: 10.1016/S0009-9236(96)90061-2. PMID 8841157
- [Background] Chaffman M, Heel RC, Brogden RN, Speight TM, Avery GS. Indapamide. A review of its pharmacodynamic properties and therapeutic efficacy in hypertension. Drugs. 1984 Sep;28(3):189-235. doi: 10.2165/00003495-198428030-00001. PMID 6489195
- [Background] Mimran A, Zambrowski JJ, Coppolani T. Indapamide in hypertension: results of a French multi-centre study in ambulant subjects. Curr Med Res Opin. 1983;8 Suppl 3:105-8. doi: 10.1185/03007998309109844. PMID 6352182
- [Background] Passeron J, Pauly N, Desprat J. International multicentre study of indapamide in the treatment of essential arterial hypertension. Postgrad Med J. 1981;57 Suppl 2:57-9. PMID 7033949
- [Background] Morledge JH. Clinical efficacy and safety of indapamide in essential hypertension. Am Heart J. 1983 Jul;106(1 Pt 2):229-32. doi: 10.1016/0002-8703(83)90121-7. PMID 6346846
- [Background] Capone P, Vukovich RA, Neiss ES, Bolton S, Reeves RL. Multicenter dose-response study of the effect of indapamide in the treatment of patients with mild to moderate hypertension. Clin Ther. 1983;5(3):305-16. PMID 6342786
- [Background] De Divitiis O, Di Somma S, Petitto M, Fazio S, Ligouri V. Indapamide and atenolol in the treatment of hypertension: double-blind comparative and combination study. Curr Med Res Opin. 1983;8(7):493-500. doi: 10.1185/03007998309109788. PMID 6354604
- [Background] Kubik MM, Coote JH. Comparison of the antihypertensive effects of indapamide and metoprolol. Postgrad Med J. 1981;57 Suppl 2:44-50. PMID 7033946
- [Background] Prisant LM; Dilacor XR/Lozol Study Group. Ambulatory blood pressure profiles in patients treated with once-daily diltiazem extended-release or indapamide alone or in combination. Am J Ther. 2000 May;7(3):177-84. doi: 10.1097/00045391-200007030-00005. PMID 11317166
- [Background] Lacourciere Y. Analysis of well-being and 24-hour blood pressure recording in a comparative study between indapamide and captopril. Am J Med. 1988 Jan 29;84(1B):47-52. PMID 3277419
- [Background] MacFadyen RJ, Lees KR, Reid JL. Differences in first dose response to angiotensin converting enzyme inhibition in congestive heart failure: a placebo controlled study. Br Heart J. 1991 Sep;66(3):206-11. doi: 10.1136/hrt.66.3.206. PMID 1657084
- [Background] Ferrari R. Angiotensin-converting enzyme inhibition in cardiovascular disease: evidence with perindopril. Expert Rev Cardiovasc Ther. 2005 Jan;3(1):15-29. doi: 10.1586/14779072.3.1.15. PMID 15723572
- [Background] Julius S, Cohn JN, Neutel J, Weber M, Turlapaty P, Shen Y, Dong V, Batchelor A, Lagast H. Antihypertensive utility of perindopril in a large, general practice-based clinical trial. J Clin Hypertens (Greenwich). 2004 Jan;6(1):10-7. doi: 10.1111/j.1524-6175.2004.02440.x. PMID 14724419
- [Background] Dahlof B, Sever PS, Poulter NR, Wedel H, Beevers DG, Caulfield M, Collins R, Kjeldsen SE, Kristinsson A, McInnes GT, Mehlsen J, Nieminen M, O'Brien E, Ostergren J; ASCOT Investigators. Prevention of cardiovascular events with an antihypertensive regimen of amlodipine adding perindopril as required versus atenolol adding bendroflumethiazide as required, in the Anglo-Scandinavian Cardiac Outcomes Trial-Blood Pressure Lowering Arm (ASCOT-BPLA): a multicentre randomised controlled trial. Lancet. 2005 Sep 10-16;366(9489):895-906. doi: 10.1016/S0140-6736(05)67185-1. PMID 16154016
- [Background] Beckett NS, Peters R, Fletcher AE, Staessen JA, Liu L, Dumitrascu D, Stoyanovsky V, Antikainen RL, Nikitin Y, Anderson C, Belhani A, Forette F, Rajkumar C, Thijs L, Banya W, Bulpitt CJ; HYVET Study Group. Treatment of hypertension in patients 80 years of age or older. N Engl J Med. 2008 May 1;358(18):1887-98. doi: 10.1056/NEJMoa0801369. Epub 2008 Mar 31. PMID 18378519
- [Background] Patel A; ADVANCE Collaborative Group; MacMahon S, Chalmers J, Neal B, Woodward M, Billot L, Harrap S, Poulter N, Marre M, Cooper M, Glasziou P, Grobbee DE, Hamet P, Heller S, Liu LS, Mancia G, Mogensen CE, Pan CY, Rodgers A, Williams B. Effects of a fixed combination of perindopril and indapamide on macrovascular and microvascular outcomes in patients with type 2 diabetes mellitus (the ADVANCE trial): a randomised controlled trial. Lancet. 2007 Sep 8;370(9590):829-40. doi: 10.1016/S0140-6736(07)61303-8. PMID 17765963
- [Background] PROGRESS Collaborative Group. Randomised trial of a perindopril-based blood-pressure-lowering regimen among 6,105 individuals with previous stroke or transient ischaemic attack. Lancet. 2001 Sep 29;358(9287):1033-41. doi: 10.1016/S0140-6736(01)06178-5. PMID 11589932
- [Background] Fox KM; EURopean trial On reduction of cardiac events with Perindopril in stable coronary Artery disease Investigators. Efficacy of perindopril in reduction of cardiovascular events among patients with stable coronary artery disease: randomised, double-blind, placebo-controlled, multicentre trial (the EUROPA study). Lancet. 2003 Sep 6;362(9386):782-8. doi: 10.1016/s0140-6736(03)14286-9. PMID 13678872
- [Background] Dahlof B, Gosse P, Gueret P, Dubourg O, de Simone G, Schmieder R, Karpov Y, Garcia-Puig J, Matos L, De Leeuw PW, Degaute JP, Magometschnigg D; PICXEL Investigators. Perindopril/indapamide combination more effective than enalapril in reducing blood pressure and left ventricular mass: the PICXEL study. J Hypertens. 2005 Nov;23(11):2063-70. doi: 10.1097/01.hjh.0000187253.35245.dc. PMID 16208150
- [Background] Mogensen CE, Viberti G, Halimi S, Ritz E, Ruilope L, Jermendy G, Widimsky J, Sareli P, Taton J, Rull J, Erdogan G, De Leeuw PW, Ribeiro A, Sanchez R, Mechmeche R, Nolan J, Sirotiakova J, Hamani A, Scheen A, Hess B, Luger A, Thomas SM; Preterax in Albuminuria Regression (PREMIER) Study Group. Effect of low-dose perindopril/indapamide on albuminuria in diabetes: preterax in albuminuria regression: PREMIER. Hypertension. 2003 May;41(5):1063-71. doi: 10.1161/01.HYP.0000064943.51878.58. Epub 2003 Mar 24. PMID 12654706
- [Background] Mourad JJ, Waeber B, Zannad F, Laville M, Duru G, Andrejak M; investigators of the STRATHE trial. Comparison of different therapeutic strategies in hypertension: a low-dose combination of perindopril/indapamide versus a sequential monotherapy or a stepped-care approach. J Hypertens. 2004 Dec;22(12):2379-86. doi: 10.1097/00004872-200412000-00021. PMID 15614033
- [Background] Sami MH. Distinctive properties of perindopril among converting enzyme inhibitors in congestive heart failure. Can J Cardiol. 1994 Nov;10 Suppl D:13D-16D. PMID 7954033
- [Background] Sonnenblick EH. Perindopril treatment for congestive heart failure. Am J Cardiol. 2001 Oct 4;88(7A):19i-27i. doi: 10.1016/s0002-9149(01)01918-x. PMID 11591357
- [Background] Macfadyen RJ, Lees KR, Reid JL. Perindopril. A review of its pharmacokinetics and clinical pharmacology. Drugs. 1990;39 Suppl 1:49-63. doi: 10.2165/00003495-199000391-00009. PMID 2407493
- [Background] O'Loughlin DC, Chu VL, Singh D. Perindopril. Heart Dis. 2000 Nov-Dec;2(6):446-55. PMID 11728296
- [Background] Hurst M, Jarvis B. Perindopril: an updated review of its use in hypertension. Drugs. 2001;61(6):867-96. doi: 10.2165/00003495-200161060-00020. PMID 11398915
- [Background] Luscher TF, Cosentino F. The classification of calcium antagonists and their selection in the treatment of hypertension. A reappraisal. Drugs. 1998 Apr;55(4):509-17. doi: 10.2165/00003495-199855040-00003. PMID 9561341
- [Background] Donnelly R. Clinical implications of indapamide sustained release 1.5 mg in hypertension. Clin Pharmacokinet. 1999;37 Suppl 1:21-32. doi: 10.2165/00003088-199937001-00004. PMID 10491730
- [Background] Mancia G, Fagard R, Narkiewicz K, Redon J, Zanchetti A, Bohm M, Christiaens T, Cifkova R, De Backer G, Dominiczak A, Galderisi M, Grobbee DE, Jaarsma T, Kirchhof P, Kjeldsen SE, Laurent S, Manolis AJ, Nilsson PM, Ruilope LM, Schmieder RE, Sirnes PA, Sleight P, Viigimaa M, Waeber B, Zannad F; Task Force Members. 2013 ESH/ESC Guidelines for the management of arterial hypertension: the Task Force for the management of arterial hypertension of the European Society of Hypertension (ESH) and of the European Society of Cardiology (ESC). J Hypertens. 2013 Jul;31(7):1281-357. doi: 10.1097/01.hjh.0000431740.32696.cc. No abstract available. PMID 23817082
- [Background] Jassim Al Khaja KA, Sequeira RP, Mathur VS. Rational pharmacotherapy of hypertension in the elderly: analysis of the choice and dosage of drugs. J Clin Pharm Ther. 2001 Feb;26(1):33-42. doi: 10.1046/j.1365-2710.2001.00324.x. PMID 11286605
- [Background] Gosse P. Perindopril/indapamide combination in the first-line treatment of hypertension and end-organ protection. Expert Rev Cardiovasc Ther. 2006 May;4(3):319-33. doi: 10.1586/14779072.4.3.319. PMID 16716093
- [Derived] Brguljan Hitij J, Gaciong Z, Simic D, Vajer P, Zelveian P, Chazova IE, Jelakovic B; Precious trial investigators. Differences in sex and age response to single pill combination based antihypertensive therapy reflecting in blood pressure and arterial stiffness. J Hypertens. 2025 Mar 1;43(3):387-396. doi: 10.1097/HJH.0000000000003901. Epub 2024 Nov 7. PMID 39445609